CLINICAL TRIAL: NCT01946347
Title: Effect of Hyperinsulinemia and Postprandial Metabolic Changes on Endothelial Function in Patients With Type 2 Diabetes Versus Healthy Subjects
Brief Title: Endothelial Function in Patients With Type 2 Diabetes Versus Healthy Subjects
Acronym: EndoPat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Responsible Party: Principal Investigator, Prof. Terezie Pelikanova, Prof.MUDr.Terezie Pelikanova DrSc., Institute for Clinical and Experimental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: G981
Record Dates: First submitted 2013-09-05; First posted 2013-09-19 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Insulin Resistance; Type 2 Diabetes
Keywords: Insulin Resistance; Hyperglycemia; Endothelial function; Oxidative stress
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with type 2 diabetes (Experimental): 30 individuals with type 2 diabetes Intervention: mixed meal, acute in vivo induced hyperinsulinemia
  Interventions: Other: mixed meal; Other: Acute in vivo induced hyperinsulinemia
- Healthy subjects (Active Comparator): 30 healthy men and women with no metabolic syndrome Intervention: mixed meal, acute in vivo induced hyperinsulinemia
  Interventions: Other: mixed meal; Other: Acute in vivo induced hyperinsulinemia

INTERVENTIONS:
Other: mixed meal — Baguette Cheese Gourmet (Crocodile:
  180g, energy 452.8 Kcal, composition: carbohydrates 49,2 g (44,55%), proteins 18,5 g (16,74%), lipids 18,8 g (38,7%), of which saturated 6,8 g, monounsaturated 6,0 g, polyunsaturated 5,0 g.
Other: Acute in vivo induced hyperinsulinemia — Hyperinsulinemic (1mU/kg/min) euglycemic clamp 3 hours long

SUMMARY:
The aim of the study is to evaluate the effect of hyperinsulinemia and postprandial changes in plasma glucose and lipids concentrations on the endothelial function together with other metabolic parameters in patients with type 2 diabetes (T2D) and in healthy subjects.

Hypothesis:

Different changes in endothelial function to acute in vivo induced hyperinsulinemia and after the meal test will be found in patients with T2D compared to healthy subjects.

A significant relationships between insulin sensitivity, selected adipokines intramyocellular fat content, hepatic fat content and high energy phosphates in soleus muscle will be documented in both groups.

DETAILED DESCRIPTION:
30 patients with T2D and 30 healthy control subjects will be examined on an outpatient basis. The following examination will be carried out in each subject after 12 hrs fasting:

* Hyperinsulinaemic euglycemic clamp study lasting 4 hours combined with indirect calorimetry and biopsy of subcutaneous adipose tissue and muscle aspiration biopsy
* Meal test:Plasma glucose, immunoreactive insulin, plasma lipids, oxidative stress markers and gastrointestinal peptides measured in response to a standard meal(at times 0´,30´,60´,120´,180´)
* At the beginning and after 120 minutes during the meal test and clamp peripheral microvascular endothelial function will be measured using EndoPat(Itamar Medical)
* Proton and phosphorus magnetic resonance spectroscopy(MRS).
* Dual Energy X-ray Absorptiometry(DXA) scanning to measure body composition.

ELIGIBILITY:
Patients with T2D:

Inclusion criteria -

1. Men and women aged 30-65 years
2. Body Mass Index in the range of 25 - 45(kg/m2)
3. Type 2 diabetes mellitus for at least one year
4. Treatment of T2D: diet or oral antidiabetic agents (stable drug therapy at least 3 months before the trial
5. The presence of metabolic syndrome - any three of the following symptoms:

   1. Abdominal obesity - waist circumference in men >102 cm, in women >88 cm
   2. Diagnosis and treatment of type 2 diabetes
   3. Raised blood pressure (BP): systolic BP > 130 mm Hg or diastolic BP >85 mm Hg, or treatment of previously diagnosed hypertension
   4. Reduced HDL cholesterol in men < 1 mmol/l, in women < 1,3 mmol/l (or treatment)
   5. Raised triglycerides > 1,7 mmol/l (or treatment)

4. HbA1c ≥ 42 a ≤100 mmol/mol

Exclusion criteria -

1. Type 1 diabetes mellitus
2. Unstable drug therapy at least 3 month before the trial
3. Pregnancy, breast feeding or trying to become pregnant
4. Alcoholism or drug use
5. Presence of other medical condition, which occurs during physical examination, laboratory tests, including pulmonary, neurological or inflammatory disease, which would be considered by the examiner to distort the consistency of data

Healthy subjects:

Inclusion criteria -

1. Men and women aged 30-65 years
2. Body Mass Index 25-45 (kg/m2)
3. Absence of metabolic syndrome - not more than any two of the following symptoms:

   1. Abdominal obesity - waist circumference in men >102 cm, in women >88 cm
   2. Diagnosis and treatment of type 2 diabetes or raised fasting plasma glucose level (FPG >5,6 mmol/l)
   3. Raised blood pressure (BP): systolic BP >130 mm Hg or diastolic BP >85 mm Hg, or treatment of previously diagnosed hypertension
   4. Reduced HDL cholesterol in men <1 mmol/l, in women <1,3 mmol/l(or treatment)
   5. Raised triglycerides > 1,7 mmol/l (or treatment)

Exclusion criteria -

1. Diabetes or impaired glucose tolerance (HbA1c ≥40 mmol/mol and/or FPG >5,6 mmol/l), diagnosed diabetes in first-line relatives
2. Pregnancy, breast feeding or trying to become pregnant
3. Alcoholism or drug use
4. Presence of other medical condition, which occurs during physical examination, laboratory tests, including pulmonary, neurological or inflammatory disease, which would be considered by the examiner to distort the consistency of data

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes of endothelial function (measured by EndoPat) | 120 minutes
  at 0 and after 120 minutes during the clamp and 120 minutes after meal ingestion

SECONDARY OUTCOMES:
Changes in gastrointestinal peptides concentrations | 180 minutes
  0, 30, 60, 120, 180 minutes after meal ingestion
Changes in oxidative stress markers | 120 minutes
  at 0 and after 120 minutes after meal ingestion
Insulin sensitivity measured as glucose disposal during clamp | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Terezie Pelikanova, Prof, MD, Principal Investigator — Diabetes Center, Institute of Clinical and Experimental Medicine
Locations (1):
- Diabetes Center, Institute of Clinical and Experimental Medicine, Prague, Czechia